CLINICAL TRIAL: NCT06980688
Title: Multicentre Single-blinded, Expertise-based RCT Comparing Haemodynamic Parameters Between Titration and Conventional Induction of General Anaesthesia With Target-controlled Infusion System in Patients Undergoing Non-cardiac Surgery
Brief Title: The PROTECT Trial: PROpofol Titration to Enhance haemodynamiC sTability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: am24DellKuster
Record Dates: First submitted 2025-05-08; First posted 2025-05-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Anesthesia
Keywords: Target-controlled infusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titration group (Experimental): Patients in the titration group undergo anaesthesia induction using a stepwise approach, where the target effect-site concentration (Cet) of propofol is incrementally increased until loss of consciousness (LOC) is achieved. Once LOC is reached, the remifentanil target concentration is elevated to mitigate the laryngeal stimulus to intubation.
  Interventions: Procedure: Propofol titration
- Conventional group (Other): Patients in the conventional group receive anaesthesia induction using a predefined high Cet of propofol, set above the typical level required to achieve loss of consciousness (LOC), aiming for rapid induction. After induction, the remifentanil target concentration is adjusted to mitigate the laryngeal stimulus of intubation.
  Interventions: Procedure: Conventional propofol induction

INTERVENTIONS:
Procedure: Propofol titration — Induction starts with propofol target-controlled Infusion (TCI) (Schnider model) at target effect-site drug concentration (Cet) 0.5-1.0 µg/mL and remifentanil TCI (Minto model) at Cet 0.5 ng/mL. If loss of consciousness (LOC) is not reached, propofol Cet is increased in 0.5-1.0 µg/mL steps. For intubation, remifentanil Cet increases up to 6.0 ng/mL.
  Arms: Titration group
Procedure: Conventional propofol induction — Induction starts with propofol TCI at Cet 4-8 µg/mL and remifentanil TCI at Cet 2.5-3.5 ng/mL.
  Arms: Conventional group

SUMMARY:
The aim of this multicentre, single-blinded, expertise-based randomised controlled trial is evaluate whether slowly increasing the dose of the anaesthetic drug propofol based on a patient's needs leads to more stable blood pressure compared to giving a standard starting dose in patients aged 55 and older undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
Propofol is a widely used anaesthetic drug known to lower blood pressure (hypotension) by relaxing blood vessels. The extent of hypotension depends on the dose and speed of propofol administration. A significant drop in blood pressure after anaesthesia is started, known as post-induction hypotension (PIH), can damage organs like the heart and kidneys, especially in older and multimorbid patients.

Target-controlled infusion (TCI) systems are commonly used to deliver anaesthetic drugs like propofol and remifentanil in a controlled way. The standard approach for starting anaesthesia (induction) is to begin with a high dose to quickly make the patient unconscious and suppress the body's response to intubation. Titration is a potentially safer alternative, where the dose is slowly increased until the patient becomes unconscious.

However, current evidence comparing the two methods is limited, especially in older patients. A small retrospective study suggested that titration improves blood pressure stability, and a survey of Swiss anaesthetists showed strong interest in this approach.

This multicentre, single-blinded, expertise-based randomised controlled trial investigates whether titration using TCI systems improves blood pressure stability in patients aged 55 and older undergoing non-cardiac surgery. The results of this trial will help to evaluate the clinical applicability and economic impact of the titration method in routine anaesthesia care and may support its future implementation into standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 55 years old
* Patients undergoing any of the following planned surgery under general anaesthesia with intubation: Ear, nose and throat, gynaecological, maxillofacial, orthopedic, plastic and reconstructive, spine, urologic, vascular (varicose vein surgery, femoral endarterectomy, peripheral bypass surgery) and visceral surgery
* Standard procedure for anaesthesia with propofol Target-Controlled Infusion (TCI) using the Schnider model and remifentanil TCI using the Minto model
* American Society of Anesthesiologists Physical Status Classification system (ASA PS) I-IV
* Body mass index (BMI) ≥18.5 or <35 kg/m2
* Signed written informed consent

Exclusion Criteria:

* Special forms of anaesthesia induction, specifically awake tracheal intubation and rapid sequence induction
* Combined anaesthesia procedures (general and regional anaesthesia combined)
* Special forms of general anaesthesia (opioid-free anaesthesia or any opioid-sparring modifications with lidocaine, magnesium, ketamine, clonidine or dexmedetomidine)
* Surgery in the prone position within the first 30 minutes
* Patients with known difficult airway
* Daily consumption of alcohol (> one unit/day) or > seven units/week
* Any regular recreational drug abuse
* Chronic use of benzodiazepines or opioids
* Allergy to propofol
* Patients with known brain pathologies, specifically seizure disorders, stroke within the past 9 months or dementia
* History of awareness
* Inability to follow procedures or insufficient knowledge in German

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Area under the mean arterial pressure threshold (AUT) | 30 min after start of induction
  The area under the mean arterial pressure (MAP)-time curve below each patient's individual baseline MAP (AUT) is measured during the first 30 minutes after the start of anaesthesia induction.

SECONDARY OUTCOMES:
Maximum Deviance (maxDev) | 30 min after start of induction
  The maximum deviation between baseline MAP and the lowest recorded MAP (maxDev) is measured during the first 30 minutes after the start of anaesthesia induction.
Use of vasoactive drugs | Up to 30 min after start of induction
  The administration of vasoactive drugs during the first 30 minutes following the start of anaesthesia induction is documented.
Use of Trendelenburg/ lithotomy positioning | Up to 30 min after start of induction
  The application of Trendelenburg/lithotomy positioning, where the patient is laid flat with the legs elevated above the head during the first 30 minutes following the start of anaesthesia induction is documented. If applied, the duration of this positioning is recorded.
Total propofol consumption | At LOC, up to 30 min after start of induction, and at skin incision
  Total propofol consumption in mg/kg is assessed at loss of consciousness (LOC), during the first 30 minutes after the start of anaesthesia induction, and at skin incision.
Neurocognitive test | before surgery, 1 and 3-5 hours after recovery of consciousness (ROC)
  To assess changes in neurocognitive performance, the validated, computerised Creyos task battery is used. Changes from baseline are used to evaluate the short-term impact of anaesthesia induction method on postoperative cognition.
Brice Interview | 3-5 hours after ROC
  To evaluate the occurrence of intraoperative awareness, the the structured and validated Brice interview is conducted postoperatively.
Time from induction start to LOC | From induction start to LOC
  The time from the start of anaesthesia induction to the onset of LOC is measured. LOC is defined by the absence of response to verbal and tactile stimuli, loss of the eyelash reflex, and no reaction to a jaw thrust manoeuvre. The time to LOC will be recorded to assess the speed of induction between different anaesthesia techniques.
Total remifentanil consumption | At LOC, up to 30 min after start of induction, and at skin incision
  Total remifentanil consumption in ug/kg is assessed at LOC, during the first 30 minutes after the start of anaesthesia induction, and at skin incision.
Time from induction start to intubation | From induction start to intubation
  The time from the start of anaesthesia induction to successful intubation is measured.
Signs of reaction to intubation | During intubation
  The occurrence of signs of reaction to intubation are recorded as yes/no. If a reaction is noted, the specific signs will be documented in free text, including but not limited to tachycardia, cough reflex, limb movement, or eye opening. This outcome will help evaluate the anaesthesia technique's ability to suppress intubation responses.
Effect-site concentration of propofol | At LOC and ROC
  The effect-site concentration (Ce) of propofol is measured at LOC and ROC.
Effect-site concentration (Ce) of remifentanil | At LOC and ROC
  The effect-site concentration (Ce) of remifentanil is measured at LOC and ROC.
Duration of MAP below threshold | Up to 30 min after start of induction
  The time that the MAP remains below 70 mmHg and 60 mmHg during the first 30 minutes following the start of anaesthesia induction is recorded.
Bispectral Index at skin incision | At skin incision
  The Bispectral Index (BIS) value at the time of skin incision as a measure of the patient's level of consciousness is recorded.
Total opioid consumption | During PACU stay
  The total opioid consumption during the post-anaesthesia care unit (PACU) stay is recorded.

OTHER OUTCOMES:
Health Economic Analysis | During the perioperative period
  This outcome focuses on the health economic analysis of the perioperative period, assessing several key cost-related metrics. These include the amount of propofol and other anaesthesia drugs used, operating theatre and PACU occupation times, staff time, and length of stay (overall and by ward type). Additionally, perioperative costs, from the hospital's perspective, are evaluated both overall and broken down by category, as well as hospitalisation costs. The aggregation of these measures will provide a comprehensive health economic outcome, reflecting the total resource utilization and associated costs in the perioperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Salome Dell-Kuster, Prof. Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (4):
- Switzerland (4):
  - Kantonsspital Baden, Baden
  - University Hospital Basel, Basel
  - Cantonal Hospital Graubünden, Chur
  - Kantonsspital Olten, soH, Olten

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data upon reasonable request
Time Frame: After publication of the data, 20 years

REFERENCES:
- [Derived] Funk S, Lohri MD, Kopp Lugli A, Schindler C, Wiencierz A, Mnich K, Schlapfer M, Gaberdiel AP, Puhan MA, Steiner LA, Gomes NV, Dell-Kuster S. The PROTECT trial: Effect of titrated versus conventional induction of general anaesthesia using a target-controlled infusion system on haemodynamics in patients undergoing non-cardiac surgery - protocol for a multicentre, expertise-based randomised controlled trial. BMJ Open. 2026 Jan 28;16(1):e110452. doi: 10.1136/bmjopen-2025-110452. PMID 41605589